CLINICAL TRIAL: NCT06502223
Title: The Impact of Microbiota and Associated Blood Tryptophan Metabolites on Pain Perception in Patients Undergoing Lumbar Disc Herniation Surgery
Brief Title: Impact of Gut Microbiota and Tryptophan Metabolites on Acute Pain in Lumbar Disc Herniation Surgery Patients
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Yunus Çelik, MD, Principal Investigator, Dokuz Eylul University
Other Study IDs: DEU-Çelik001
Record Dates: First submitted 2024-06-28; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Microbial Substitution; Tryptophan Metabolism Alterations; Postoperative Pain, Acute
Keywords: Microbiota; Tryptophan; Picolinic Acid; Kynurenic Acid; Xanthurenic Acid; Quinolinic Acid; Acute Pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pain Perception in Patients Undergoing Lumbar Disc Herniation Surgery — Analyze tryptophan metabolites (picolinic acid, 3- Hydroxykynurenine, anthranilic acid, kynurenine, quinolinic acid, kynurenic acid, xanthurenic acid). Concurrent VAS pain assessments were conducted, and correlations between tryptophan metabolites and VAS were evaluated.
  Other Names: Microbiota and Associated Blood Tryptophan Metabolites on

SUMMARY:
It is well-established that the gut microbiota plays a crucial role in various pain mechanisms, including visceral pain, inflammatory pain, headache, neuropathic pain, and opioid tolerance. Changes in the gut microbiome can alter pain perception. In our study, The investigator investigated the effects of microbiota alterations and the associated tryptophan metabolites on acute pain using the Visual Analog Scale (VAS).

DETAILED DESCRIPTION:
The study included patients aged 18 and above undergoing lumbar disc herniation surgery. Blood samples were collected preoperatively, at 8 hours, and at 24 hours postoperatively to analyze tryptophan metabolites (picolinic acid, 3- Hydroxykynurenine, anthranilic acid, kynurenine, quinolinic acid, kynurenic acid, xanthurenic acid). Concurrent VAS pain assessments were conducted, and correlations between tryptophan metabolites and VAS were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar disc herniation surgery at Dokuz Eylül University Hospital.
* Patients who have read and consented to the informed consent form for the study.
* Age 18 years or older.
* Surgery duration exceeding 2 hours.

Exclusion Criteria:

* Patients are unwilling to participate in the study.
* Surgery duration less than 2 hours.
* Patients under the age of 18.
* Patients with a history of abdominal surgery.
* Patients who received antibiotic therapy for intestinal pathology within the last 3 weeks.
* Patients with known abdominal pathologies suspected to alter the microbial flora (e.g., Crohn's disease, ulcerative colitis, celiac disease).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our study includes 37 lumbar disc herniation (LDH) surgeries performed in Dokuz Eylül University Faculty of Medicine Central Operating Rooms Brain and Nerve Surgery Hall. For the blood samples in which the investigators evaluated tryptophan metabolites; 2 mL of blood was used from the blood samples taken during routine surgery preparation for the patients and from the routine blood samples taken in the postoperative period, and no additional invasive intervention was performed.
  Concurrently with each blood draw, the patient's VAS score, the nature of the pain, and vital signs were recorded. Patient records, clinical histories, examination findings, and relevant laboratory results were electronically recorded.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Tryptophan metabolites (Picolinic Acid) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  2 mL of blood was used from the blood samples taken during routine surgery preparation for the patients and from the routine blood samples taken in the postoperative period, and no additional invasive intervention was performed. The investigator elucidated the relationship between picolinic acid and its variations due to microbiota alterations with VAS in acute pain. Preoperative, postoperative, 8th-hour, and 24th-hour blood samples were routinely collected from patients, with 2 mL of sample material used each time. After the necessary centrifugation processes, the relevant laboratory team analyzed the picolinic acid levels (ng/mL).
Tryptophan metabolites (3-Hydroxykynurenine) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  2 mL of blood was used from the blood samples taken during routine surgery preparation for the patients and from the routine blood samples taken in the postoperative period, and no additional invasive intervention was performed. The investigator elucidated the relationship between 3-Hydroxykynurenine and its variations due to microbiota alterations with VAS in acute pain. Preoperative, postoperative 8th-hour, and 24th-hour blood samples were routinely collected from patients, with 2 mL of sample material used each time. After the necessary centrifugation processes, the relevant laboratory team analyzed the 3-Hydroxykynurenine levels(ng/mL).
Tryptophan metabolites (Anthranilic Acid) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  2 mL of blood was used from the blood samples taken during routine surgery preparation for the patients and from the routine blood samples taken in the postoperative period, and no additional invasive intervention was performed. The investigator elucidated the relationship between anthranilic acid and its variations due to microbiota alterations with VAS in acute pain. Preoperative, postoperative, 8th-hour, and 24th-hour blood samples were routinely collected from patients, with 2 mL of sample material used each time. The relevant laboratory team measured the anthranilic acid levels (ng/mL) following the required centrifugation procedures.
Tryptophan metabolites (Kynurenine) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  2 mL of blood was used from the blood samples taken during routine surgery preparation for the patients and from the routine blood samples taken in the postoperative period, and no additional invasive intervention was performed. The investigator elucidated the relationship between kynurenine and its variations due to microbiota alterations with VAS in acute pain. Preoperative, postoperative, 8th-hour, and 24th-hour blood samples were routinely collected from patients, with 2 mL of sample material used each time. After the necessary centrifugation processes, the relevant laboratory team analyzed the kynurenine levels (ng/mL).
Tryptophan metabolites (Quinolinic Acid) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  2 mL of blood was used from the blood samples taken during routine surgery preparation for the patients and from the routine blood samples taken in the postoperative period, and no additional invasive intervention was performed. The investigator elucidated the relationship between quinolinic acid and its variations due to microbiota alterations with VAS in acute pain. Preoperative, postoperative, 8th-hour, and 24th-hour blood samples were routinely collected from patients, with 2 mL of sample material used each time. After the necessary centrifugation processes, the relevant laboratory team analyzed the quinolinic acid levels (ng/mL).
Tryptophan metabolites (Kynurenic Acid) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  2 mL of blood was used from the blood samples taken during routine surgery preparation for the patients and from the routine blood samples taken in the postoperative period, and no additional invasive intervention was performed. The investigator elucidated the relationship between kynurenic acid and its variations due to microbiota alterations with VAS in acute pain. Preoperative, postoperative, 8th-hour, and 24th-hour blood samples were routinely collected from patients, with 2 mL of sample material used each time. After the necessary centrifugation processes, the relevant laboratory team analyzed the kynurenic acid levels (ng/mL).
Tryptophan metabolites (Xanthurenic Acid) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  2 mL of blood was used from the blood samples taken during routine surgery preparation for the patients and from the routine blood samples taken in the postoperative period, and no additional invasive intervention was performed. The investigator elucidated the relationship between xanthurenic acid and its variations due to microbiota alterations with VAS in acute pain. Preoperative, postoperative, 8th-hour, and 24th-hour blood samples were routinely collected from patients, with 2 mL of sample material used each time. After the necessary centrifugation processes, the relevant laboratory team analyzed the xanthurenic acid levels (ng/mL).
Visual Analog Scale | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  In VAS assessment, patients are typically asked to choose a value between "0, no pain" and "10, the worst imaginable pain." VAS is an 11-point scale (ranging from 0 to 10) that allows patients to numerically express the intensity of their pain. Blood samples were planned and collected from patients during the preoperative evaluation, at the 8th postoperative hour, and at the 24th postoperative hour, adhering to clinical routines for these procedures. Concurrently with each blood draw, the patient's VAS score, the nature of the pain, and vital signs were recorded.

SECONDARY OUTCOMES:
Systolic Blood Pressure (mmHg) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  The study measured the systolic blood pressure (mmHg) of patients at specified time points.The patients' systolic blood pressure data were recorded simultaneously with the blood samples taken during routine surgery preparation and at the 8th and 24th hours postoperatively.
Diastolic Blood Pressure (mmHg) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  The study measured the diastolic blood pressure (mmHg) of patients at specified time points.The patients' diastolic blood pressure data were recorded simultaneously with the blood samples taken during routine surgery preparation and at the 8th and 24th hours postoperatively.
Pulse Rate (beats per minute) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  The study measured patients' pulse rate (beats per minute) at specified time points.The patients' pulse data were recorded simultaneously with the blood samples taken during routine surgery preparation and at the 8th and 24th hours postoperatively.
Respiratory Rate (breaths per minute) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  The study measured the respiratory rate (breaths per minute) of patients at specified time points.
  The patients' respiratory rate data were recorded simultaneously with the blood samples taken during routine surgery preparation and at the 8th and 24th hours postoperatively.
Oxygen Saturation (%) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  The study measured patients' oxygen saturation (%) at specified time points.The patients' oxygen saturation data were recorded simultaneously with the blood samples taken during routine surgery preparation and at the 8th and 24th hours postoperatively.
Nature of Postoperative Pain Assessed by the McGill Pain Questionnaire (MPQ) | Preoperative: Before surgery; Postoperative 8th-hour: 8 hours after surgery;Postoperative 24th-hour: 24 hours after surgery
  The McGill Pain Questionnaire (MPQ) was used to evaluate and categorize the nature of pain. The study assessed the nature and quality of acute postoperative pain using the McGill Pain Questionnaire (MPQ) at specified time points. Although all of the patients' pain was acute postoperative pain, the pain qualities were recorded simultaneously, taking into account the differences in pain qualities. The MPQ was used to evaluate and categorize the nature of pain. The MPQ includes descriptors of pain which are categorized into sensory, affective, evaluative, and miscellaneous dimensions. Each descriptor is rated on an intensity scale of 0 (none) to 3 (severe), and scores are summed to provide an overall pain score. Higher scores indicate worse pain.
Comorbidity Assessment in Relation to Pain and Tryptophan Metabolites | Preoperative anamnesis process: Prior to surgery, during patient assessment, Follow-up: Through study completion, an average of 1 year
  The study recorded patients' comorbidities, specifically those identified during the preoperative anamnesis process, and evaluated their potential impact on the nature of pain and tryptophan metabolites. Comorbidities identified as exclusion criteria, particularly those believed to affect intestinal microbiota and related to abdominal conditions, were also considered. Patients' comorbidities identified during the preoperative anamnesis process were meticulously documented to assess their influence on pain characteristics and tryptophan metabolites. Additionally, comorbidities identified as exclusion criteria due to their potential to alter intestinal microbiota and their association with abdominal conditions were thoroughly evaluated.
Anesthesia induction drugs | During anesthesia procedure
  Although standardization of drugs used in anesthesia is difficult, standardization of induction drugs was partially achieved because the investigators chose a single surgery group. The investigators recorded all of this data during anesthesia applications.
Anesthesia duration and surgery times | During surgery
  Our study detailedly recorded the duration of anesthesia and surgery. To ensure a certain level of standardization, we included only lumbar disc surgery, which is considered sterile. Additionally, surgeries shorter than a specified duration were excluded as they might not provide significant metabolic changes. These durations were carefully recorded throughout the entire surgery and anesthesia period. The investigators accepted these durations as one of the elimination criteria due to their potential impact on pain and physiological mechanisms.
Age of Investigator | Preoperative: During the preoperative anamnesis process
  The investigator's age was recorded during the preoperative anamnesis process to understand its influence on the study variables.
Weight of Investigator | Preoperative: During the preoperative anamnesis process
  The weight of the investigator was recorded during the preoperative anesthesia process to understand its influence on the study variables.
Height of Investigator | Preoperative: During the preoperative anamnesis process
  The height of the investigator was recorded during the preoperative anamnesis process to understand its influence on the study variables.
Body Mass Index (BMI) of Investigator | Preoperative: During the preoperative anamnesis process
  The Body Mass Index (BMI) of the investigator was calculated from recorded height (in meters) and weight (in kilograms) during the preoperative anamnesis process to understand its influence on the study variables.BMI values are reported in units of kg/m².
Gender of Investigator | Preoperative: During the preoperative anamnesis process
  The gender of the investigator was recorded during the preoperative anamnesis process to understand its influence on the study variables.

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Celik, M.D., Study Chair — Dokuz Eylül University Hospital, Faculty of Medicine
Locations (1):
- Yunu Çelik, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The investigators do not see any harm in sharing the data of our study to contribute to other studies and meta-analyses. The investigators received our informed consent, but the investigators made such a choice because the investigators doubted that it would be public.

REFERENCES:
- [Derived] Celik Y, Aksu H, Gunenc FS, Kalemci O, Kizmazoglu C, Keskinoglu P. Association between circulating tryptophan metabolites and postoperative pain intensity in lumbar disc herniation surgery: An observational study. Medicine (Baltimore). 2025 Aug 1;104(31):e43704. doi: 10.1097/MD.0000000000043704. PMID 40760513

DOCUMENTS (3):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT06502223/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT06502223/SAP_001.pdf
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/23/NCT06502223/ICF_002.pdf